CLINICAL TRIAL: NCT01587131
Title: Phase I, Open Label Study of a DNA Vaccine's Ability to Increase the Immune Response to the Trivalent Seasonal Influenza Vaccine in the Elderly
Brief Title: DNA-based Influenza Vaccine in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2011:131
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2013-01

CONDITIONS: Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases
Keywords: Universal Influenza; Intradermal DNA-Based Vaccine; Senior; Electroporation; H1; Influenza; FVH1
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1- DNA prime DNA boost (Experimental): 0.9 mg of FVH1 vaccine delivered ID followed by electroporation on Day 0, Week 15 and Week 27
  Interventions: Biological: FVH1 - a DNA-based influenza vaccine
- Group 2 - DNA prime Seasonal Vaccine boost (Experimental): 0.9 mg FVH1 vaccine delivered ID followed by electroporation on Day 0 and Trivalent Seasonal Influenza Vaccine delivered IM on Week 15
  Interventions: Biological: FVH1 - a DNA-based influenza vaccine
- Group 3 - sWFI prime Seasonal Vaccine boost (Placebo Comparator): 100 microliters of sterile water for injection delivered ID followed by electroporation on Day 0 and Trivalent Seasonal Influenza Vaccine delivered IM on Week 15
  Interventions: Biological: FVH1 - a DNA-based influenza vaccine

INTERVENTIONS:
Biological: FVH1 - a DNA-based influenza vaccine — 0.9 mg FVH1 vaccine

SUMMARY:
The purpose of this study is to determine whether FVH1, a DNA-based influenza vaccine, will be safe and generally well tolerated in healthy elderly adult volunteers and will result in greater immunogenicity when used to prime the immune response to a dose of a trivalent inactivated seasonal vaccine.

DETAILED DESCRIPTION:
The use of DNA plasmids containing genes that express viral antigens may be a promising way to formulate a vaccine that can effectively prevent infection and disease caused by the H1N1 influenza virus. Plasmid vectors are simple to construct and are easy to manufacture at a relatively low cost. Vaccination with plasmids that express influenza proteins should induce the development of serum antibodies and might also induce significant quantities of secretory IgA antibodies and/or CMI. The DNA sequences included in the vaccine could also result in the proliferation of T lymphocytes that could broaden the effectiveness of the vaccine to include variant strains of H1N1 with antigenically modified HA (i.e., drifted strains).

Electroporation (EP) is a technology in which a transmembrane electrical field is applied to increase the permeability of cell membranes to create microscopic pathways (pores) and thereby enhance the uptake of drugs, vaccines, or other agents into target cells. Their presence allows macromolecules, ions, and water to pass from one side of the membrane to the other. The presence of a constant field influences the kinetics of directional translocation of the macromolecular plasmid, such that the plasmid delivery in vivo has been sufficient to achieve physiological levels of secreted proteins. ID injection of a plasmid followed by EP has been used very successfully to deliver therapeutic genes that encode for a variety of hormones, cytokines, or enzymes in a variety of species. EP is currently being used in humans to deliver cancer vaccines and therapeutics as well as in gene therapy. The expression levels are increased by as much as 3 orders of magnitude over plasmid injection alone.

The use of EP via the CELLECTRA® device should increase the expression of H1N1 influenza virus genes in the study vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines;
* Adults of either gender ≥ 65 years of age at entry;
* Healthy subjects, as judged by the Qualified Investigator based on medical history, physical examination, and normal results of an electrocardiogram (ECG), complete blood count (CBC), serum chemistries, and urinalysis done up to 4 weeks prior to enrollment and administration of vaccine or placebo by ID/EP;
* Current non-smoker (for 3 months prior to vaccine study);
* Willing to forego any other influenza vaccination during the study;
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site (excluding inhaled and eye drop-containing corticosteroids) or the use of other immunosuppressive agents. All other corticosteroids must be discontinued ≥ 4 weeks prior to Day 1 of study vaccine administration;
* Administration of any blood product within 3 months of enrollment;
* Subjects with contraindications to influenza vaccination other than egg allergy (such as a history of Guillain-Barre Syndrome after receiving influenza vaccine);
* Administration of any vaccine within 6 weeks of enrollment; subjects may not receive any licensed seasonal influenza vaccine during the study unless they have been assigned to a study group receiving the seasonal vaccine;
* Participation in a study with an investigational compound or device within 4 weeks of signing informed consent;
* Subjects with cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
* Subjects with a history of seizures (unless seizure free for 5 years);
* Subjects with tattoos, scars, or active lesions/rashes within 2 cm of the site of vaccination + EP;
* Subjects with any implanted heart leads;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
* Prisoner subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a DNA-based influenza vaccine composed of a combination of two different H1 HA plasmids administered ID followed by electroporation in healthy elderly adult subjects | Day 0 through Month 12
  Frequency and severity of local and systemic reactogenicity signs and symptoms, adverse events and serious adverse events

SECONDARY OUTCOMES:
Humoral and cellular immune responses | Day 0 through Month 12
  Magnitude and frequency of antibody and cell mediated immune response to influenza proteins

CONTACTS AND LOCATIONS:
Overall Officials: Gary Kobinger, PhD, Principal Investigator — National Microbiology & University of Manitoba; Trina Racine, PhD, Study Director — National Microbiology Laboratory, Canada
Locations (1):
- MS Building Health Sciences Centre, Winnipeg, Manitoba, Canada